CLINICAL TRIAL: NCT05522530
Title: Cross-cultural Adaptation, Reliability, Validity and Viability of the Mini Bestest in Balance Disorders Upon Admission or Readmission to Vestibular Rehabilitation in the Autonomous City of Buenos Aires: Validation Study Protocol
Brief Title: Cross-cultural Adaptation and Validity of Mini Bestest in Balance Disorders in the Autonomous City of Buenos Aires: Validation Study Protocol
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital de Rehabilitacion Manuel Rocca (Other)
Responsible Party: Principal Investigator, Marcos Ceferino Gabriel Valdez, Physical Therapist, Hospital de Rehabilitacion Manuel Rocca
Other Study IDs: 5884
Record Dates: First submitted 2022-08-28; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Vestibular Disease; Peripheral Vestibular Disorder
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment scale — Evaluation scale to carry out its cross-cultural adaptation and study its validity

SUMMARY:
The objective of this study is to carry out the cross-cultural adaptation of the Mini BESTest (a balance assessment scale) into Argentine Spanish, as well as to study its validation in patients with peripheral vestibular disorders in the autonomous city of Buenos Aires.

ELIGIBILITY:
Inclusion Criteria:

* Subjects >18 years of age,
* With vestibular alterations of peripheral etiology, within the second year of evolution
* Time of evolution of symptoms ≤ 2 years
* Independent walking with or without walking assistance device
* Who are at the beginning of a VR program
* No diagnoses of psychiatric disorders or cognitive impairment,
* Sign the informed consent

Exclusion Criteria:

* Who have suffered amputation in one of their lower limbs,
* History of neurological pathologies (stroke, multiple sclerosis, neuromuscular disease)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with peripheral vestibular disorders
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Mini BESTest | 1 hour
  Assessment scale of postural balance

CONTACTS AND LOCATIONS:
Locations (1):
- Marcos Ceferino Gabriel Valdez, Almagro, Buenos Aires F.D., Argentina